CLINICAL TRIAL: NCT06236308
Title: A Randomized, Phase 1 Dose Finding Study of TTAX03 for the Treatment of Lumbosacral Facet Joint Pain
Brief Title: TTAX03 for the Treatment of Lumbosacral Facet Joint Pain
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was stopped due to reprioritization for active studies
Sponsor: BioTissue Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTAX03-CR007
Record Dates: First submitted 2023-11-06; First posted 2024-02-01 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Facet Joint Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TTAX03 10mg (Experimental): TTAX03 is a sterile, lyophilized and micronized particulate human AM and UC product manufactured using aseptic processing followed by terminal sterilization by gamma irradiation in compliance with current Good Tissue Practices (cGTP) and current Good Manufacturing Practices (cGMP) to preserve extracellular matrices and growth factors/cytokines therein without any living cells. 10 mg of TTAX03 in a 0.5 mL solution of sterile, preservative-free 0.9% NaCl (saline).
  Interventions: Biological: TTAX03 10mg
- TTAX03 25mg (Experimental): TTAX03 is a sterile, lyophilized and micronized particulate human AM and UC product manufactured using aseptic processing followed by terminal sterilization by gamma irradiation in compliance with current Good Tissue Practices (cGTP) and current Good Manufacturing Practices (cGMP) to preserve extracellular matrices and growth factors/cytokines therein without any living cells. 25 mg TTAX03 in a 0.5 mL saline solution; or 0.5 mL of saline alone.
  Interventions: Biological: TTAX03 25mg
- Saline Control (Placebo Comparator): 0.5 mL of saline alone
  Interventions: Biological: Placebo Comparator: Control Saline

INTERVENTIONS:
Biological: TTAX03 10mg — TTAX03 is a sterile, lyophilized and micronized particulate human AM and UC product manufactured using aseptic techniques followed by terminal sterilization by gamma-irradiation in compliance with Current Good Tissue Practices (CGTP) and Current Good Manufacturing Practices (CGMP) to preserve extracellular matrices and growth factors/cytokines therein without any living cells.
  Arms: TTAX03 10mg
Biological: TTAX03 25mg — TTAX03 is a sterile, lyophilized and micronized particulate human AM and UC product manufactured using aseptic techniques followed by terminal sterilization by gamma-irradiation in compliance with Current Good Tissue Practices (CGTP) and Current Good Manufacturing Practices (CGMP) to preserve extracellular matrices and growth factors/cytokines therein without any living cells.
  Arms: TTAX03 25mg
Biological: Placebo Comparator: Control Saline — 2 mL Sterile, preservative free 0.9% NaCl
  Arms: Saline Control

SUMMARY:
This is a pilot study examining the safety and efficacy of a single intra-articular (IA) injection of TTAX03 per joint to relieve severe spinal facet joint (FJ) pain and improve function in subjects with facet joint pain (FJP) in the lumbosacral region. The design is randomized, double blinded, placebo controlled and dose-group sequential.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, placebo-controlled, double-blinded dose ranging study design with two dose escalation cohorts to be conducted at three sites in the USA. The primary objective is to examine the safety of FJ IA injections with the test article. The fundamental framework for the number of subjects and dose escalation decisions is modeled on the widely utilized phase 1 "3+3" dose escalation design.

A second objective is to examine the efficacy of two doses of TTAX03. The efficacy null hypothesis (HO) is that one administration of TTAX03, introduced into each of two or four joints (at one or two levels) by IA injection, will have no more benefit with respect to pain relief and improved function than an equal volume of placebo (sterile saline). The alternate hypothesis (HA) is that TTAX03 will provide a clinically meaningful reduction in pain and improvement in function compared to placebo.

An exploratory objective is to examine the potential benefit in terms of reduced need for narcotic pain relief, radiofrequency ablation, or surgical procedures for relief of LBP.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent
2. Women of childbearing potential (those who are not premenarchal, not surgically sterilized [hysterectomy or bilateral oophorectomy], or not post-menopausal) may participate in the study if they meet all of the following conditions:

   * they are not breast feeding
   * they have a negative serum pregnancy test at screening
   * they agree to undertake a serum pregnancy test at screening, at 3 months, and upon exiting the study
   * they do not intend to become pregnant during the study
   * they are using adequate birth control methods and they agree to continue using those methods for the duration of the study

   Adequate birth control methods are defined as: hormonal-topical, oral, implantable or injectable contraceptives; mechanical-spermicide in conjunction with a barrier such as a condom or diaphragm; IUD; or, surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, she must agree to use an adequate birth control method as described above for the remainder of the study.

   NOTE: Women who have had a bilateral tubal ligation are not considered to have been surgically sterilized and must agree to the conditions as specified above.

   Post-menopausal is defined as no menstrual period for at least one year.
3. ≥ 35 and ≤ 85 years of age
4. BMI <40 kg/m2
5. Clinical suspicion of painful OA of the facet joint(s) in 1 to 4 lumbosacral joints (within 1 - 2 levels) of greater than 3 months duration.
6. Evidence of OA of the facet in the lumbosacral region on MRI or X-ray within 3 months (e.g., joint space narrowing, the presence of osteophytes and/or subchondral cysts, articular process hypertrophy, subchondral bone sclerosis, articular and subarticular erosions).
7. NRS score for "worst pain in the past 24 hrs" ≥ 5, using the first NRS value collected in the screening period.
8. History of having attempted a regimen of conservative care, including physical therapy for ≥ 3 months.
9. Positive response to two diagnostic MBB, defined as ≥ 80% reduction in pain, at any time within 1 hour, assessed at 1 hour, as self-reported by the subject, following each diagnostic block.
10. White blood count ≥ 4,500 /uL, absolute neutrophil count (ANC) > 1,000 / uL, platelet count ≥ 75,000 /uL, Hgb ≥ 10 g/dL
11. Normal prothrombin time (PT) and partial thromboplastin time (PTT).
12. Hemoglobin A1c (HbA1c) ≤ 8%
13. Adequate hepatic function (AST/ALT ≤ 1.5 × ULN, total bilirubin ≤ 1.2 × ULN)
14. Adequate renal function (eGFR ≥ 60 mL/min/1.73 m2)
15. Currently insufficient pain relief from acetaminophen, NSAIDs or other non-opioid analgesic medications.

Exclusion Criteria:

1. Lactation or pregnancy
2. Cardiovascular instability as indicated by any of the following identified at screening and verified at least once during the initial screening visit: uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic >100 mm Hg), uncontrolled arrhythmia or unstable angina pectoris.
3. Cognitive impairment, mental illness, neuroses or untreated depression that would preclude understanding or reliably completing the patient reported outcome measures
4. History within the past 12 months of gastrointestinal bleeding, myocardial infarction, chronic renal failure, hepatic fibrosis, chronic obstructive pulmonary disease, or hospitalization other than for elective procedures
5. Non-ambulatory, bedridden, or with active fibromyalgia or central pain syndrome
6. Hypoesthesia, paresthesia, or allodynia in either foot or leg
7. Facet OA pain involving more than two levels (i.e., > 4 FJs)
8. Use of > 30 morphine milligram equivalents (MME) per day (see Study Guide)
9. Score ≥ 21 on the Beck Depression Inventory (BDI)
10. Allergy to any local anesthetic agents
11. Any of the following conditions:

    1. Local (spine) or systemic infection
    2. Tumor in the spine
    3. Acute (< 3 months duration) vertebral fracture

    e. Systemic inflammatory disorder f. Radicular syndrome g. Cauda equina syndrome h. Ankylosing spondylitis i. Any arthritis not considered osteoarthritis, such as reactive, rheumatoid, psoriatic or enteropathic arthritis j. History of other autoimmune disease or Crohn's disease
12. Progressive neurological condition such as Parkinson's, Alzheimer's, Lou Gehrig's disease, etc.
13. Clinical characteristics suggestive of discogenic pain (i.e., chronic low back pain that subsides in supine position but aggravated after long-time sitting or standing, radicular pain)
14. Radiologic evidence and radicular pain indicating symptomatic herniated disc
15. Sacroiliac joint pain or symptomatic nerve root impingement (neurogenic claudication) related to spinal stenosis
16. Evidence of dynamic listhesis, or fixed listhesis >10 mm accompanied by intermittent claudication or spinal stenosis
17. Corticosteroid injections within 1 month of screening if injected into the lumbar spine remote from the index facet joints, or within 3 months of screening if injected into the index facet joints, or radiofrequency ablation treatment at any level in the lumbar spine within 6 months of screening for similar symptoms
18. Prior surgery at the involved levels, including "failed back syndrome"
19. History of spinal osteonecrosis, osteoporotic fracture, fracture around the index facet joint(s) within the past 3 years, or pars interarticularis defect
20. Compensable disability or work injury, ongoing or anticipated litigation related to back injury
21. Sickle cell disease
22. Erythrocyte sedimentation rate (ESR) >40mm/hr
23. Use of systemic immunosuppressive medications within past 6 months, including chronic systemic corticosteroids, chemotherapy, or history of organ transplant (kidney, heart, lung)
24. Concurrent treatment, or treatment in the past 6 months, with any investigational agent
25. Severe concurrent illness which, in the view of the investigator, would interfere with this 12-month study

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Physical, functional and physiological responses to the intervention, as well as unanticipated events | 12-weeks post baseline
  Proportion of subjects with developing or worsening abnormalities on focused motor, sensory and reflex neurological exams;
  - and - Changes from baseline in blood chemistries, hematology, serum immunoglobulins, urinalysis, and markers of inflammation

SECONDARY OUTCOMES:
NRS pain score | At the end of 12, 26, 39, and 52 weeks following treatment, compared to placebo
  >/ 30% reduction in the NRS pain score
PROMIS-29 | At the end of 12, 26, 39, and 52 weeks following treatment, compared to placebo
  Improvement by >/ 5 points on the PROMIS-29
NRS pain score | At the end of 1, 4, 8, and 12 weeks following treatment, compared to placebo
  Change from baseline in NRS value
PROMIS-29 | At the end of 12, 26, 39 and 52 weeks, compared to placebo
  Change from baseline in PROMIS-29
ODI score | At the end of 12, 26, 39 and 52 weeks, compared to placebo
  Change from baseline in ODI score
PGIC | At the end of 12, 26, 39 and 52 weeks, compared to placebo
  Change from baseline in PGIC

OTHER OUTCOMES:
Frequency and amount of narcotic use, radiofrequency ablation and surgical intervention | Following treatment with TTAX03 or placebo after 12 weeks
  Exploratory- To characterize the need for alternative treatment